CLINICAL TRIAL: NCT03812848
Title: Implementation of Clinical Pharmacist-led Inpatient Anticoagulation Stewardship Program in An Egyptian Tertiary Care Hospital
Brief Title: Clinical Pharmacist-led Inpatient Anticoagulation Stewardship Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Heba Mohamed El-Bosily, Clinical Pharmacist, Ain Shams University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 165
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Deep Vein Thrombosis; Atrial Fibrillation; Mitral Valve Disease
Keywords: anticoagulation; stewardship program; anticoagulants; clinical pharmacist; heparin; warfarin
MeSH Terms: conditions — Venous Thrombosis; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Quasi experimental study (separate sample pre-test post-test design)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre program implementation (No Intervention): All hospitalized patients on therapeutic anticoagulant medication during the pre-implementation period of the anticoagulation stewardship program.
- Post program implementation (Experimental): All hospitalized patients on therapeutic anticoagulant medication during the post-implementation period of the anticoagulation stewardship program.
  Interventions: Other: Anticoagulation Stewardship Program

INTERVENTIONS:
Other: Anticoagulation Stewardship Program — A clinical-pharmacist led anticoagulation stewardship program that includes:
  1. Warfarin monitoring and dosing protocol. 1a.Warfarin initial dosing algorithm. 1b.Recommended International normalized ration (INR) target and duration of Warfarin therapy by indication.
  1c.Warfarin dosage adjustment algorithms.
  1d.Management of high INR values. 2-Heparin weight-based protocol. 3-Perioperative anticoagulation use protocol. 4-Policies that address baseline and ongoing laboratory monitoring for anticoagulants.
  5-Protocol for Heparin Induced Thrombocytopenia(HIT) management. 6-Anticoagulation reversal protocol. 7-Booklet for anticoagulant drugs and all of previously prepared protocols. 8-Education programs regarding anticoagulation's therapy for health care team dealing with anticoagulation and patients.
  Arms: Post program implementation

SUMMARY:
This study aims at evaluating the implementation of clinical-pharmacist-led anticoagulation stewardship program in Egyptian tertiary hospital to promote a culture of safety around anticoagulants.

DETAILED DESCRIPTION:
One of the high-alert medication categories that may cause significant patient harm if not used correctly is anticoagulants. It is not clear if medication errors are more common with this category in specific compared to other medication categories, but the ramifications of a medication error with the use of anticoagulation agents is without a doubt detrimental to the patient's health and more serious than most of other drug categories.

This prospective study evaluates the impact of implementing an anticoagulation stewardship program, led by clinical pharmacists, on anticoagulation therapy outcomes during patient hospitalization by the percent of medication errors reduction, percent of adverse drug events reduction, and percent of evidence-based guidelines compliance improvement.

ELIGIBILITY:
Inclusion Criteria:

All hospitalized patients on therapeutic anticoagulant medication during their hospitalization period.

Exclusion Criteria:

1. Patients whose age is less than 18 years old.
2. Patients who were admitted for less than 24 hours for patient on parenteral anticoagulants and less than 48 hours for patient on warfarin.
3. Patients already admitted for bleeding or thrombosis.
4. Malignancy patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Percent of medication errors change | one year and half
  Detect the medication error according to (National Coordinating Council for Medication Errors Reporting and Prevention NCC MERP) Index for Categorizing Medication Errors using NCC MERP Index for Categorizing Medication Errors Algorithm.
percent of adverse drug events change | one year and half
  Detect bleeding and thrombotic-related adverse drug events
Percent of evidence-based guidelines compliance improvement | one year and half
  Detect health care providers' adherence to evidence-based guidelines for anticoagulation therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
It is not clear according to the clinical research guidelines at Faculty of Pharmacy, Ain Shams University.

REFERENCES:
- [Background] Broussard M, Bass PF 3rd, Arnold CL, McLarty JW, Bocchini JA Jr. Preprinted order sets as a safety intervention in pediatric sedation. J Pediatr. 2009 Jun;154(6):865-8. doi: 10.1016/j.jpeds.2008.12.022. Epub 2009 Feb 1. PMID 19181332
- [Background] Burnett AE, Trujillo TC. The future of inpatient anticoagulation management. J Thromb Thrombolysis. 2013 Apr;35(3):375-86. doi: 10.1007/s11239-013-0892-1. PMID 23417781
- [Background] Dreijer AR, Kruip MJ, Diepstraten J, Polinder S, Brouwer R, Leebeek FW, Vulto AG, van den Bemt PM. Antithrombotic stewardship: a multidisciplinary team approach towards improving antithrombotic therapy outcomes during and after hospitalisation: a study protocol. BMJ Open. 2016 Dec 20;6(12):e011537. doi: 10.1136/bmjopen-2016-011537. PMID 27998897
- [Background] Fanikos J, Stapinski C, Koo S, Kucher N, Tsilimingras K, Goldhaber SZ. Medication errors associated with anticoagulant therapy in the hospital. Am J Cardiol. 2004 Aug 15;94(4):532-5. doi: 10.1016/j.amjcard.2004.04.075. PMID 15325949
- [Background] Garcia DA, Baglin TP, Weitz JI, Samama MM. Parenteral anticoagulants: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e24S-e43S. doi: 10.1378/chest.11-2291. PMID 22315264
- [Background] Goldspiel B, Hoffman JM, Griffith NL, Goodin S, DeChristoforo R, Montello CM, Chase JL, Bartel S, Patel JT. ASHP guidelines on preventing medication errors with chemotherapy and biotherapy. Am J Health Syst Pharm. 2015 Apr 15;72(8):e6-e35. doi: 10.2146/sp150001. No abstract available. PMID 25825193
- [Background] Levinson, D. R., & General, I. (2010). Adverse events in hospitals: national incidence among Medicare beneficiaries. Department of Health and Human Services Office of the Inspector General. Retrieved from https://oig.hhs.gov/oei/reports/oei-06-09-00090.pdf
- [Background] Levy JH, Spyropoulos AC, Samama CM, Douketis J. Direct oral anticoagulants: new drugs and new concepts. JACC Cardiovasc Interv. 2014 Dec;7(12):1333-51. doi: 10.1016/j.jcin.2014.06.014. PMID 25523529
- [Background] Hug BL, Witkowski DJ, Sox CM, Keohane CA, Seger DL, Yoon C, Matheny ME, Bates DW. Adverse drug event rates in six community hospitals and the potential impact of computerized physician order entry for prevention. J Gen Intern Med. 2010 Jan;25(1):31-8. doi: 10.1007/s11606-009-1141-3. Epub 2009 Nov 6. PMID 19894081
- [Background] Lysogorski MC, Hassan AK, Lampkin SJ, Geisler R. The impact of pharmacy monitoring and intervention in patients receiving intravenous heparin. Int J Clin Pharm. 2017 Aug;39(4):844-850. doi: 10.1007/s11096-017-0482-y. Epub 2017 May 15. PMID 28508323
- [Background] Padron M, Miyares MA. Development of an anticoagulation stewardship program at a large tertiary care academic institution. J Pharm Pract. 2015 Feb;28(1):93-8. doi: 10.1177/0897190013514091. Epub 2013 Dec 10. PMID 24326411
- [Background] Reardon DP, Atay JK, Ashley SW, Churchill WW, Berliner N, Connors JM. Implementation of a Hemostatic and Antithrombotic Stewardship program. J Thromb Thrombolysis. 2015 Oct;40(3):379-82. doi: 10.1007/s11239-015-1189-3. PMID 25669625
- [Background] Rose, A. (Ed.). (2015). Anticoagulation Management. Cham: Springer International Publishing. https://doi.org/10.1007/978-3-319-22602-6
- [Background] Sharma M, Krishnamurthy M, Snyder R, Mauro J. Reducing Error in Anticoagulant Dosing via Multidisciplinary Team Rounding at Point of Care. Clin Pract. 2017 Apr 20;7(2):953. doi: 10.4081/cp.2017.953. eCollection 2017 Apr 6. PMID 28484587
- [Background] U.S. Department of Health and Human Services, Office of Disease Prevention and Health Promotion. (2014). Anticoagulants. In National Action Plan for Adverse Drug Event Prevention.
- [Background] World Health organization, W. H., & others. (2016). Medication Errors: Technical Series on Safer Primary Care ISBN 978-92-4-151164-3. Retrieved from http://apps.who.int/iris/bitstream/10665/252275/1/9789241511650-eng.pdf
- [Background] Wychowski MK, Ruscio CI, Kouides PA, Sham RL. The scope and value of an anticoagulation stewardship program at a community teaching hospital. J Thromb Thrombolysis. 2017 Apr;43(3):380-386. doi: 10.1007/s11239-016-1455-z. PMID 27878507
- See also: Institute for Safe Medication Practices. (2010). ISMP's Guidelines for Standard Order Sets. — http://www.ismp.org/guidelines/standard-order-sets
- See also: Institute for Safe Medication Practices. (2014). ISMP list of High-Alert Medications — http://www.ismp.org/recommendations/high-alert-medications-acute-list
- See also: Institute for Safe Medication Practices (ISMP) Monitoring FDA MedWatch Reports. (2015, September). Quarter Watch (Q 3-4) 2014. Institute for Safe Medication Practices (ISMP). — http://www.ismp.org/quarterwatch
- See also: Institute for Safe Medication Practices (ISMP) ,Quarter Watch (Q4): monitoring FDA MedWatch Reports. (2017, July). Quarter Watch Q4 2016. Retrieved July 13, 2017, from http://www.ismp.org/QuarterWatch/ — http://www.ismp.org/quarterwatch?combine=&field_date_posted_value=&page=3
- See also: NCCMERP. (2014, July 18). Types of Medication Errors [Text]. — http://www.nccmerp.org/types-medication-errors